CLINICAL TRIAL: NCT06480136
Title: An Exploratory Clinical Study of SHR-A1921 Combined With Adebrelimab in the Treatment of Advanced NSCLC Who Failed the Previous Standard First-line Treatment
Brief Title: SHR-A1921 Combined With Adebrelimab in the Treatment of Advanced NSCLC Who Failed the Previous Standard First-line Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of clinical research center, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024LY0534
Record Dates: First submitted 2024-06-25; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: NSCLC
Keywords: Trop-2 ADC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): SHR-A1921+adebrelimab
  Interventions: Drug: SHR-A1921 injection and adebrelimab injection

INTERVENTIONS:
Drug: SHR-A1921 injection and adebrelimab injection — The Treatment group receive SHR-A1921 injection combined with adebrelimab injection

SUMMARY:
This is a Phase II clinical study to evaluate the efficacy and safety of SHR-A1921 conbined with adebrelimab in advanced NSCLC who failed the previous first-line standard therapy. Subjects in this study were treated with SHR-A1921 in combination with adebrelimab until disease progression, intolerable toxicity occurs, informed consent is withdrawn, or other conditions requiring termination of medication, whichever occurred first. The maximum treatment time of adebrelimab is 35 cycles or 2 years (whichever comes first), and subjects can continue to be treated with SHR-A1921 until disease progression, intolerable toxicity occurs, informed consent is withdrawn, or other conditions requiring termination of medication. Primary objective of this study was to evaluate the efficacy of SHR-A1921 combined with adebrelimab in advanced NSCLC who failed the previous first-line standard therapy. Secondary objective of this study was to evaluate the safety of SHR-A1921 combined with adebrelimab in advanced NSCLC who failed the previous first-line standard therapy; Exploratory objective of this study was to evaluate the biomarker changes during treatment with SHR-A1921 combined with adebrelimab in patients with advanced NSCLC who failed the previous first-line standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to join in this study, signed informed consent, good adherence, can cooperate with the follow-up;
2. Age 18-75 years old, both genders;
3. Patients with histologically or cytologically confirmed advanced or metastatic NSCLC（Advanced stage is defined as stage IIIb-IV according to the 8th edition of the IASLC TNM staging criteria), and no longer suitable for radical surgery or radiotherapy combined with chemotherapy；
4. Participants with nonsquamous tumors were required to have available genetic testing to confirm without EGFR, ALK, or ROS1 driver mutations;
5. Disease progression after prior immunization (PD-1/L1 antibody)or combined with platinum-based chemotherapy;
6. At least one measurable lesion that met RECIST v1.1 criteria;
7. ECOG Performance Status of 0-1;
8. Must have life-expectancy of ≥ 12 weeks;
9. Adequate function of marrow and major organs meets the following requirements：

   1. Blood routine (no blood transfusion or granulocyte colony-stimulating factor therapy within 14 days before examination)：ANC≥1.5×109/L；PLT≥75×109/L；Hb≥90 g/L;
   2. Liver function (no hepatoprotective drugs within 7 days before the examination): ALT and AST≤3 × ULN (liver metastasis≤5.0 × ULN); TBIL≤1.5 × ULN（Gilbert's syndrome subjects: TBIL≤3mg/dL）;
   3. Renal function:Cr≤1.5 × ULN or creatinine clearance ≥60 mL / min (Cockcroft-Gault formula)；
   4. Coagulation: INR or PT≤1.5×ULN，APTT≤1.5×ULN；
   5. Cardiac ultrasound: LVEF≥50%;
10. Female patients of childbearing age or male patients whose partner was a female of childbearing age had to consent to use a highly effective method of contraception for the duration of the study and for 6 months after the last dose of study drug; and have no plans to have children or to donate sperm or eggs, Childbearing age female patients who were not surgically sterilized had to undergo a serum pregnancy test with a negative result within 7 days before starting study treatment.；

Exclusion Criteria:

1. Previous receipt of any drug containing a topoisomerase I inhibitor drug, including antibody-drug conjugates;
2. Previous receipt of TROP2-targeted therapy;
3. Grade 3 or above immune-related adverse events occurred during previous immunotherapy, such as immune-related interstitial lung disease, immune-related myocarditis, immune hepatitis, etc.
4. More than 10% of the tumor tissue was histologically or cytologically confirmed as small-cell lung cancer, neuroendocrine carcinoma, carcinosarcoma;
5. Untreated brain metastasis, or associated with meningeal metastasis, spinal cord compression, etc. Patients who had received previous treatment for brain metastases (radiotherapy or surgery) were eligible for enrollment if they had been stable for at least 4 weeks as confirmed by imaging and had been free of systemic hormone therapy (at a dose of >10 mg per day of prednisone or the equivalent) for more than 2 weeks and were asymptomatic;
6. Spinal cord compression that could not be cured by surgery and/or radiotherapy;
7. Patients with uncontrolled cancer-related pain as judged by the investigator;
8. Patients with symptomatic pleural effusion, pericardial effusion, or ascites requiring drainage or those who had undergone therapeutic drainage of serous effusion within 2 weeks before the administration of the study drug;
9. Patients who received anti-tumor therapy such as chemotherapy within 4 weeks before the first dose of medication, or received lung field radiotherapy >30Gy within 6 months before the first dose of medication;
10. Major organ surgery or major trauma within 4 weeks before the first dose of the study drug;
11. Other malignant tumors occurred within 5 years before the first treatment;
12. Patients with a history of interstitial lung disease such as idiopathic pulmonary fibrosis or imaging examination at screening that suspected interstitial pneumonia or could not rule out interstitial pneumonia;
13. Active pulmonary tuberculosis infection was detected by medical history or CT examination within 1 year before enrolment;
14. Severe infection within 4 weeks before the first dose of medication;
15. Have serious cardiovascular and cerebrovascular diseases;
16. Patients with clinically significant bleeding symptoms within 3 months before the first study medication;
17. Arterial/venous thrombotic events within 6 months before the first dose of study medication;
18. Hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg); A history of hypertensive crisis or hypertensive encephalopathy;
19. Refractory nausea, vomiting, chronic gastrointestinal diseases, etc.
20. Subjects with active, known or suspected autoimmune disease (including Hiv-Positive), or a history of organ transplantation;
21. Presence of active hepatitis B or C;
22. A live or attenuated vaccine was administered within 4 weeks before the first dose of the study drug;
23. The adverse reactions of antineoplastic therapy have not recovered to NCI-CTCAE v5.0 grade ≤ 1;
24. A history of severe allergic reaction with other monoclonal antibodies or have allergic reactions to any component of SHR-A1921 and adbelimumab;
25. According to the investigator's judgment, there are other factors that may affect the results of the study or lead to the forced termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental diseases) requiring combined treatment, serious laboratory test abnormalities, accompanied by family or social factors, which will affect the safety of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Screening up to study completion, an average of 2 year
  Objective response rate represents the proportion of patients showing a predefined level of tumor shrinkage or disappearance in response to treatment.

SECONDARY OUTCOMES:
Progression-free Survival | Screening up to study completion, an average of 2 year
  Progression-free survival measures the length of time during and after treatment that a patient lives with the disease. without it progressing.
Duration of response | Screening up to study completion, an average of 2 year
  Duration of response refers to the length of time during which a patient's tumor remains in remission or shows a positive response to treatment.
Overall Survival | Screening up to study completion, an average of 2 year
  Overall survival measures the length of time from the start of treatment until death from any cause, indicating the effectiveness of the treatment in prolonging patients' lives.
Disease control rate | Screening up to study completion, an average of 2 year
  Disease control rate refers to the proportion of patients whose tumors shrink or stabilize for a certain period of time, including complete response (CR), partial response (PR), and stable disease (SD) cases.

IPD SHARING:
Plan to Share IPD: Yes
Public article